CLINICAL TRIAL: NCT06393829
Title: Implementation of an Early Mobilization Program in Cardiovascular Units
Brief Title: Early Mobilization in Cardiovascular Units
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Interdisciplinary Research in Rehabilitation of Greater Montreal (Other)
Collaborators: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Sara Ahmed, Prof., Centre for Interdisciplinary Research in Rehabilitation of Greater Montreal
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-4090
Record Dates: First submitted 2024-03-18; First posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Cardiovascular Diseases
Keywords: Early mobilization program; cardiovascular; Level of mobility
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: The proposed project will follow the steps of the Knowledge-to-Action framework (KTA) [7]. The KTA is a process model that provides practical guidance in planning and implementing research evidence into practice [8]. It is comprised of a Knowledge Creation Funnel and an Action Cycle. Our project will follow the steps of the Action Cycle from adapting to the local context through evaluating outcomes with a concern for sustaining knowledge use.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- pre-implementation (No Intervention): The proportion of patients mobilized pre-intervention period
- Implementation (Experimental): The proportion of patients mobilized during the intervention implementation period
  Interventions: Behavioral: Applying the Early Mobilization Program
- Post-implementation (No Intervention): The proportion of patients mobilized post-intervention period

INTERVENTIONS:
Behavioral: Applying the Early Mobilization Program — A mobilization intervention based on the level of function (LOF) ( i.e. patients should be assessed for mobilization status within 24 hours of admission; mobilization should occur at least three times a day, and mobility should be progressive and scaled, tailored to the patient's abilities); The frequency of patient mobilization (primary outcome) will be assessed 20 weeks before implementation, during the 20 weeks of implementation and 20 weeks after the end of implementation (60 weeks in total).
  Arms: Implementation

SUMMARY:
Insufficient mobility contributes to functional decline in hospitalized cardiac patients. Early mobilization programs were shown to improve functional status, increase the likelihood of home discharges, and reduce the length of stay [1]. Therefore, there is a need to adapt and implement early mobilization programs in Quebec hospitals. The overall goal of this study is to adapt and implement an early mobilization program in the Cardiovascular units of the Jewish General Hospital (JGH).

DETAILED DESCRIPTION:
Background: Insufficient mobility contributes to functional decline in cardiovascular units. Early mobilization programs were shown to improve functional status, increase the likelihood of home discharges, and reduce the length of stay [1]. One example is the Level of Function (LOF) Mobility Scale implemented in the Cardiovascular units at the Jewish General Hospital, an academic tertiary care centre in Montreal, Quebec [2]. Despite evidence supporting the benefits of early mobilization programs, hospitalized individuals in cardiovascular units spend most of the day in bed [1-6]. Therefore, there is a need to adapt and implement early mobilization programs in Quebec hospitals. This project is research nested in a quality improvement initiative for the Jewish General Hospital Cardiovascular units.

Objectives: 1) Adapt an early mobilization program in a hospital setting; 2) Develop strategies to overcome individual and organizational barriers to implementing an early mobilization program; 3) Assess the reach, acceptability, and fidelity of implementing an early mobilization program; and 4) Assess the program's impact on patients and the organization.

Methods: A 3-phase study using an iterative participative approach. Phase 1: a qualitative design to adapt an early mobilization program. Phase 2: mixed methods repeated measures design to assess barriers and facilitators to implementing the program and develop implementation strategies.

Phase 3: An interrupted time series design to assess the implementation and the impact of the program.

Expected contribution: Early mobilization programs in the Cardiovascular units can improve the quality of care provided to these patients and promote further clinician-researcher partnerships, contributing to improved uptake of best practices in this clinical context.

ELIGIBILITY:
Inclusion Criteria:

* All healthcare professionals working in the cardiovascular unit at the Jewish General Hospital.
* All patients admitted to the cardiovascular unit at the Jewish General Hospital.

Exclusion Criteria:

* Patients who don't speak English or French.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Number of implementation strategies developed to overcome the identified individual and organizational barriers and leverage the facilitators to implement an early mobilization program in this hospital setting. | 3 months
  Investigators will develop strategies to overcome identified barriers and leverage the facilitators to implement the early mobilization program using data obtained from a mixed methods repeated measures design, including:
  A) Shadowing: an observational grid will be developed, including frequency of mobilization, length of mobilization activity, Health care professionals (HCPs) performing mobilization intervention, type of mobilization intervention, patient and caregiver acceptance and reaction, environmental barriers, available equipment, communication strategies among HCPs, reporting of mobilization interventions in the medical charts, clinicians' comment and observers' impressions and thoughts.
  B) HCPs will be invited to respond to a survey and participate in a focus group to assess perceived barriers and facilitators to early mobilization.
  C) Patients and caregivers will participate in a focus group to better understand barriers and facilitators to early mobilization.
Number of patients mobilized divided by the total number of admitted patients during the evaluation period. | 3 months
  Reach of the early mobilization program among patients will be measured with the following indicator: the number of patients mobilized (defined as the patient not being in bed during direct observation) divided by the total number of admitted patients during the evaluation period.
Number of Patients refused being mobilized compared to number of admited patients during the evaluation period. | 3 months
  Acceptability of the early mobilization program among patients will be measured with the refusal rate of being mobilized using the site's administrative data and a file audit that will include a form developed for this purpose.
Number of days between admission and the development of a mobilization plan, between admission and first mobilization and number of patients with at least 3 mobilizations per day per week. | 3 months
  Fidelity of intervention among HCPs will be measured with the following indicators:
  * Number of days between admission and the development of a mobilization plan
  * Number of days between admission and first mobilization
  * Number of patients with at least 3 mobilizations per day per week.
Change in mobility levels during the unit's stay. | 3 months
  Change in in mobility levels according to the LOF mobility scaleoccurring during the unit's stay.
Change in number of Pressure ulcers occurance in the unit during the evaluation period. | 3 months
  Change in Pressure ulcers rate in the unit during the evaluation period.
Number of fall incidents occurring in the unit' during the evaluation period. | 3 months
  Change in rate of falls occurring in the unit' during the evaluation period.
Change in Length of stay | 3 months
  Change in organizational outcomes measured by change in number of days the patient stay in the hospital.
Number of patients discharged to home versus number discharged to an institutional care. | 3 months
  Number of patients discharged to home versus number discharged to an institutional care used to evaluate the Effect of early monbilization on the discharge destination (home or institutional care).

CONTACTS AND LOCATIONS:
Overall Officials: Sara Ahmed, Principal Investigator — McGill univeristy
Locations (1):
- Centre for Interdisciplinary Research in Rehabilitation of Greater Montreal/Centre de rech interdisciplinaire en réadaptation du Montréal métropolitain, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
The research assistant will de-identify the participants by generating a random code using a statistical method. The research team will extract and transfer the data using a password-protected Excel spreadsheet where modification is traceable. The private information (participant personal information, i.e., name, birth date) will be coded (unique code for each participant).
  The data capturing, coding, and analysis will be conducted on a password-protected computer at Constance Lethbridge Rehabilitation center connected to a secured server.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data, informed consent forms, and questionnaires completed by patients and health care professionals will be stored at the Constance Lethbridge Rehabilitation Center on the institution's secure server by the researcher in charge of the study for ten years after the end of the project after which they will be permanently destroyed.
Access Criteria: A research assistant and a statistician will analyze and code the de-identified research data under the supervision of Sara Ahmed and Diana Zidarov, the two principal investigators. These people will have access to the data for analytical purposes.

REFERENCES:
- [Background] Anekwe DE, Biswas S, Bussieres A, Spahija J. Early rehabilitation reduces the likelihood of developing intensive care unit-acquired weakness: a systematic review and meta-analysis. Physiotherapy. 2020 Jun;107:1-10. doi: 10.1016/j.physio.2019.12.004. Epub 2019 Dec 19. PMID 32135387
- [Background] Dima D, Valiquette J, Berube-Dufour J, Goldfarb M. Level of function mobility scale for nurse-driven early mobilisation in people with acute cardiovascular disease. J Clin Nurs. 2020 Mar;29(5-6):778-784. doi: 10.1111/jocn.15124. Epub 2019 Dec 18. PMID 31793086
- [Background] Castro-Avila AC, Seron P, Fan E, Gaete M, Mickan S. Effect of Early Rehabilitation during Intensive Care Unit Stay on Functional Status: Systematic Review and Meta-Analysis. PLoS One. 2015 Jul 1;10(7):e0130722. doi: 10.1371/journal.pone.0130722. eCollection 2015. PMID 26132803
- [Background] TEAM Study Investigators; Hodgson C, Bellomo R, Berney S, Bailey M, Buhr H, Denehy L, Harrold M, Higgins A, Presneill J, Saxena M, Skinner E, Young P, Webb S. Early mobilization and recovery in mechanically ventilated patients in the ICU: a bi-national, multi-centre, prospective cohort study. Crit Care. 2015 Feb 26;19(1):81. doi: 10.1186/s13054-015-0765-4. PMID 25715872
- [Background] Zanni JM, Korupolu R, Fan E, Pradhan P, Janjua K, Palmer JB, Brower RG, Needham DM. Rehabilitation therapy and outcomes in acute respiratory failure: an observational pilot project. J Crit Care. 2010 Jun;25(2):254-62. doi: 10.1016/j.jcrc.2009.10.010. Epub 2009 Nov 26. PMID 19942399
- [Background] Dubb R, Nydahl P, Hermes C, Schwabbauer N, Toonstra A, Parker AM, Kaltwasser A, Needham DM. Barriers and Strategies for Early Mobilization of Patients in Intensive Care Units. Ann Am Thorac Soc. 2016 May;13(5):724-30. doi: 10.1513/AnnalsATS.201509-586CME. PMID 27144796
- [Background] Graham ID, Logan J, Harrison MB, Straus SE, Tetroe J, Caswell W, Robinson N. Lost in knowledge translation: time for a map? J Contin Educ Health Prof. 2006 Winter;26(1):13-24. doi: 10.1002/chp.47. PMID 16557505
- [Background] Nilsen P. Making sense of implementation theories, models and frameworks. Implement Sci. 2015 Apr 21;10:53. doi: 10.1186/s13012-015-0242-0. PMID 25895742